CLINICAL TRIAL: NCT03308084
Title: Effects of Intraoperative Local Steroid Utilization in a Single-Level Minimally Invasive Transforaminal Lumbar Interbody Fusion
Brief Title: Use of Local Intraoperative Steroid in MIS TLIF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Kern Singh, Professor, Department of Orthopaedic Surgery, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 15052003
Record Dates: First submitted 2017-10-05; First posted 2017-10-12 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Dysphasia
Keywords: transforaminal lumbar interbody fusion, methylprednisolone
MeSH Terms: conditions — Aphasia | interventions — Methylprednisolone; Dexamethasone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local Depomedrol plus IV dexamethasone (Active Comparator): Local intraoperative application of methylprednisolone (Depomedrol) plus standard systemic (IV) dexamethasone
  Interventions: Drug: Methylprednisolone; Drug: Dexamethasone
- IV dexamethasone (Placebo Comparator): Standard systemic (IV) dexamethasone only
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Methylprednisolone — Application of 80mg Depomedrol (methylprednisolone acetate) suspension into the transforaminal space prior to incision closure
  Arms: Local Depomedrol plus IV dexamethasone
Drug: Dexamethasone — Administration of 10mg Dexamethasone IV intraoperatively

SUMMARY:
The purpose of this study is to determine if the frequency and duration of postoperative pain are improved in participants receiving a local steroid injection (methylprednisolone) plus a systemic (intravenous (IV, by vein)) steroid (dexamethasone) when compared to those receiving a systemic (IV) steroid (dexamethasone) alone. Both of these steroid injections are already currently used at Rush and are considered standard of practice. It is well established that steroids have an anti-inflammatory (decreased swelling) effect on the soft tissue and it is routinely used in many types of surgery, but it is not known whether two steroids are better than one. The medications provided in this study are approved by the Food and Drug Administration (FDA).

DETAILED DESCRIPTION:
Postoperative pain is a well-known complication following minimally invasive transforaminal lumbar interbody fusion (MIS TLIF). It has been found that up to 40% of lumbar spinal patients will have either recurrent or persistent postoperative pain. Several studies have demonstrated reduced patient reported pain scores following steroid administration. However, few studies have investigated intraoperative local injection of corticosteroid at the surgical site in an effort to reduce the incidence and duration of postoperative pain for MIS TLIF patients.

The purpose of this study is to determine if the incidence and duration of postoperative pain is improved in participants receiving a local injection of methylprednisolone with systemic dexamethasone when compared to those receiving the usual systemic dexamethasone undergoing MIS TLIF.

The investigators hypothesize that participants undergoing MIS TLIF who receive local methylprednisolone along with the systemic dexamethasone will have:

1. Reduced incidence and duration of postoperative pain compared to participants receiving only systemic dexamethasone.
2. Shorter hospital stay compared to participants receiving only systemic dexamethasone.
3. Better short- and long-term outcomes compared to participants receiving only systemic dexamethasone

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a primary 1- to 2-level MIS TLIF
* Diagnosis: myelopathy, radiculopathy, myeloradiculopathy, stenosis, herniated nucleus pulposus, degenerative disc disease, spondylosis, osteophytic complexes, and foraminal stenosis
* Patients able to provide informed consent

Exclusion Criteria:

* Allergies or other contraindications to medicines in the protocol including:

  (a) Existing history of gastrointestinal bleeding
* Current Smokers
* Lumbar spine trauma
* Bilateral cages
* Lack of consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2015-11-13 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2019-05-03 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain | 2 years postoperative
  Change in Visual Analogue Scale Back and Leg score from preoperative value will be assessed

SECONDARY OUTCOMES:
Physical Functioning | 2 years postoperative
  Patient-Reported Outcomes Measurement Information System score as compared to preoperative value
Disability | 2 years postoperative
  Oswestry Disability Index score as compared to preoperative score
General health status | 2 years postoperative
  Short Form-12 Survey scores as compared to preoperative value
Narcotic Consumption | 1 week postoperative
  The total amount of narcotic use for each subject will be recorded. Dosages of narcotics will be converted to morphine equivalents
Length of Stay | 1 week postoperative
  The number of hours of hospitalization from entering the recovery room (time zero) until patient meets discharge criteria.
Intra-operative adverse events | day of surgery
  Blood loss, length of surgery, procedural details, complications
Post-operative adverse events | 1 week postoperative
  Post-operative nausea and vomiting, Gastro-esophageal reflux, Ileus, Venous thromboembolic events, Respiratory depression/airway compromise, Renal insufficiency, Wound Complications, Admission to the ICU

CONTACTS AND LOCATIONS:
Overall Officials: Kern Singh, MD, Principal Investigator — Rush University Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schizas C, Tzinieris N, Tsiridis E, Kosmopoulos V. Minimally invasive versus open transforaminal lumbar interbody fusion: evaluating initial experience. Int Orthop. 2009 Dec;33(6):1683-8. doi: 10.1007/s00264-008-0687-8. Epub 2008 Nov 21. PMID 19023571
- [Background] McGirt MJ, Parker SL, Lerner J, Engelhart L, Knight T, Wang MY. Comparative analysis of perioperative surgical site infection after minimally invasive versus open posterior/transforaminal lumbar interbody fusion: analysis of hospital billing and discharge data from 5170 patients. J Neurosurg Spine. 2011 Jun;14(6):771-8. doi: 10.3171/2011.1.SPINE10571. Epub 2011 Mar 18. PMID 21417699
- [Background] Ranguis SC, Li D, Webster AC. Perioperative epidural steroids for lumbar spine surgery in degenerative spinal disease. A review. J Neurosurg Spine. 2010 Dec;13(6):745-57. doi: 10.3171/2010.6.SPINE09796. PMID 21121754
- [Background] Jamjoom BA, Jamjoom AB. Efficacy of intraoperative epidural steroids in lumbar discectomy: a systematic review. BMC Musculoskelet Disord. 2014 May 5;15:146. doi: 10.1186/1471-2474-15-146. PMID 24885519
- [Background] Debi R, Halperin N, Mirovsky Y. Local application of steroids following lumbar discectomy. J Spinal Disord Tech. 2002 Aug;15(4):273-6. doi: 10.1097/00024720-200208000-00002. PMID 12177541
- [Derived] Haws BE, Khechen B, Patel DV, Bawa MS, Ahn J, Bohl DD, Mayo BC, Massel DH, Guntin JA, Cardinal KL, Singh K. Impact of local steroid application in a minimally invasive transforaminal lumbar interbody fusion: results of a prospective, randomized, single-blind trial. J Neurosurg Spine. 2018 Nov 9;30(2):222-227. doi: 10.3171/2018.7.SPINE18584. Print 2019 Feb 1. PMID 30497132